CLINICAL TRIAL: NCT01365221
Title: SWITCH 600/60: The Effect of Reloading Prasugrel in a Patient Who Has Already Received a Loading Dose (LD) of Clopidogrel
Brief Title: The Effect of Reloading Prasugrel in a Patient Who Has Already Received a Loading Dose (LD) of Clopidogrel
Acronym: SWITCH 600/60
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWITCH 600/60
Record Dates: First submitted 2011-05-11; First posted 2011-06-03 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute Coronary Syndrome; Clopidogrel; Prasugrel
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients who have received loading dose of clopidogrel (Experimental)
  Interventions: Drug: Prasugrel
- Patients who have not received loading dose of clopidogrel (Active Comparator)
  Interventions: Drug: Prasugrel

INTERVENTIONS:
Drug: Prasugrel — Patients who have received 600 mg loading dose of clopidogrel will receive a reloading dose of 60 mg prasugrel
  Arms: Patients who have received loading dose of clopidogrel
Drug: Prasugrel — Patients who have not received a loading dose of clopidogrel will receive a 60 mg loading dose of prasugrel.
  Arms: Patients who have not received loading dose of clopidogrel

SUMMARY:
The primary objective of this study is to compare platelet reactivity between patients receiving a loading dose of clopidogrel and a reloading dose of prasugrel to patients receiving only a loading dose of prasugrel.

DETAILED DESCRIPTION:
This is a prospective, open-label, non-randomized trial of approximately 260 patients with Acute Coronary Syndrome (ACS) undergoing percutaneous coronary intervention (PCI). In order to compare platelet reactivity, as assessed by the VerifyNow P2Y12 assay, we plan to recruit two study groups of interest:

1. Patients who have already received a 600 mg loading dose (LD) of clopidogrel in preparation for PCI will receive a loading dose of 60 mg of prasugrel.
2. Patients who have not received a LD of clopidogrel will receive a 60 mg LD of prasugrel prior to PCI.

A subset of 40 patients from each study group (80 patients total) will undergo additional platelet reactivity testing with the vasodilator stimulated phosphoprotein (VASP) assay.All patients will be followed throughout the duration of the hospital stay.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 18 or older, of both genders
2. Presenting with an ACS, defined as at least two of the following:

   Symptoms consistent with myocardial ischemia; ST segment elevation or depression of at least 1 mm in 2 or more contiguous leads on EKG; Cardiac troponin I level above the upper limit of normal.
3. An initial invasive strategy (e.g. early angiography) is planned.
4. No contraindications to prasugrel therapy.

Exclusion Criteria:

1. Known allergies to aspirin, clopidogrel, or prasugrel.
2. Patient known to be pregnant or lactating.
3. Patient with known history of bleeding diathesis, or currently active bleeding.
4. Platelet count <100,000/mm3 at the time of enrollment.
5. Hematocrit <25% at the time of enrollment.
6. On warfarin therapy at the time of PCI, or patient likely to require warfarin therapy post-PCI.
7. Received fibrinolytics within the past 48 hours.
8. Received a glycoprotein IIb/IIIa inhibitor within the past 48 hours, or if a strategy for PCI involving a glycoprotein IIb/IIIa inhibitor is planned.
9. Taking maintenance thienopyridine therapy in the previous 7 days.
10. Known blood transfusion within the preceding 10 days.
11. Patients treated with non-steroidal anti-inflammatory drugs (NSAIDS) within the previous 5 days.
12. Patients with known chronic liver disease.
13. Age greater than 75 years.
14. Body weight less than 60 kg.
15. History of stroke or transient ischemic attack.
16. Surgery planned within 1 month.
17. Patient likely to require coronary artery bypass grafting.
18. Any significant medical condition that, in the investigator's opinion, may interfere with the patient's optimal participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
The primary objective is to compare platelet reactivity, as assessed by the VerifyNow P2Y12 assay, between patients receiving a loading dose of clopidogrel and a reloading dose of prasugrel to patients receiving only a loading dose of prasugrel. | Average hospital stay is 24-48 hours.

SECONDARY OUTCOMES:
The secondary objective of this study is to describe rates of bleeding events associated with a loading dose of prasugrel in patients who have already received a loading dose of clopidogrel. | Average hospital stay is 24-48 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Ron Waksman, MD, Principal Investigator — Medstar Health Research Institute
Locations (4):
- United States (4):
  - The Heart Center, Huntsville, Alabama
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Sinai Center for Thrombosis Research, Baltimore, Maryland
  - Saint Luke's Hospital, Kansas City, Missouri

REFERENCES:
- [Result] Lhermusier T, Lipinski MJ, Drenning D, Marso S, Chen F, Torguson R, Waksman R. Switching patients from clopidogrel to prasugrel in acute coronary syndrome: impact of the clopidogrel loading dose on platelet reactivity. J Interv Cardiol. 2014 Aug;27(4):365-72. doi: 10.1111/joic.12139. Epub 2014 Jul 19. PMID 25041356